CLINICAL TRIAL: NCT06153550
Title: The Benefit of Preparation in Respiratory Physiotherapy Before a Sternotomy in the Context of Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN522021/CHUSTE
Record Dates: First submitted 2023-11-23; First posted 2023-12-01 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-11

CONDITIONS: Sternotomy
Keywords: Cardiac surgery; Sternotomy; respiration; Spirometry; pulse oximetry
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who have sternotomy: Patients who have sternotomy wll be included. They will have preparation in Respiratory Physiotherapy before sternotomy.
  Interventions: Other: preparation in Respiratory Physiotherapy

INTERVENTIONS:
Other: preparation in Respiratory Physiotherapy — preparation in Respiratory Physiotherapy consist to:
  * 3 sessions per week with the physiotherapist
  * spirometry and pulse oximetry test 3 weeks before surgery, the day before surgery and the day after surgery.

SUMMARY:
The sternotomy has some influence on the respiratory system after cardiac surgery, considerably increasing the risk of perioperative and postoperative breathing.

There is respiratory preparation before cardiac surgery using local physiotherapeutic guidelines.

DETAILED DESCRIPTION:
The aim of the study is to have a quantification of this preparation spirometry: before starting the preparation and at the end of the preparation (right before surgery) by comparing the spirometric and pulse oximetry information. The prospective study will be conducted on 25 patients, who will be selected consecutively without randomization.

ELIGIBILITY:
Inclusion Criteria:

* Patient with indication of cardiac surgery

Exclusion Criteria:

* Patient with a Body Mass Index (BMI) > 30
* Restrictive patient
* Obstructive patient
* Asthmatic
* Chronic Obstructive Pulmonary Disease (COPD)
* History of pulmonary fibrosis, tuberculosis
* Coronary patients with stenosis of the common trunk.
* Emergency and lifesaving surgeries
* History of thoracic trauma
* Severe kyphotic patients
* History of radiotherapy
* Patients with neuromuscular disease
* Patients with thoracic cage involvement (pectus excavatum, post thoracic surgery)
* Patients with emphysema
* Patients with dilated bronchi

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patient with indication of cardiac surgery will be included.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2021-11-10 (Actual)

PRIMARY OUTCOMES:
Analysis of the evolution of the pulmonary function by Forced spirometry. | 3 weeks before, the day before and the day after surgery.
  Measured by spirometry and pulse oximetry results.

SECONDARY OUTCOMES:
Analysis of the evolution of the pulmonary function by Resistance | 3 weeks before, the day before and the day after surgery.
  Measured by spirometry and pulse oximetry results.
Analysis of the evolution of the pulmonary function by Lung volumes | 3 weeks before, the day before and the day after surgery.
  Measured by spirometry and pulse oximetry results.
Analysis of the evolution of the pulmonary function by Dissemination capacity, | 3 weeks before, the day before and the day after surgery.
  Measured by spirometry and pulse oximetry results.
Analysis of the evolution of the pulmonary function by Flow / volume curves | 3 weeks before, the day before and the day after surgery.
  Measured by spirometry and pulse oximetry results.
Analysis of the evolution of the pulmonary function by Peripheral saturation | 3 weeks before, the day before and the day after surgery.
  Measured by spirometry and pulse oximetry results.

CONTACTS AND LOCATIONS:
Overall Officials: Andranik PETROSYAN, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No